CLINICAL TRIAL: NCT04636359
Title: Dongzhimen Hospital Affiliated to Beijing University of Chinese Medicine
Brief Title: Study the Effect of Acupuncture on Migraine Patient Without Aura Via Functional Magnetic Resonance Imaging.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yi Ren, Deputy director of Neurology, Beijing University of Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BeijingUCM-KWu
Record Dates: First submitted 2020-11-04; First posted 2020-11-19 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Migraine Without Aura
Keywords: Acupuncture; Functional magnetic resonance imaging
MeSH Terms: conditions — Migraine without Aura

STUDY DESIGN:
Intervention Model Description: Two experimental groups with different condition receive identical intervention, with control group as baseline for comparison.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long term course of migraine patient without aura (Experimental): Patients in this group have the history of migraine without aura more than 5 years.
  Interventions: Behavioral: Acupuncture stimulation
- Short term course of migraine patient without aura (Experimental): Patients in this group have the history of migraine without aura equal or less than 5 years.
  Interventions: Behavioral: Acupuncture stimulation

INTERVENTIONS:
Behavioral: Acupuncture stimulation — The intervention is about acupuncture treatment, which has 4 weeks acupoint stimulation and the frequency is 30 minutes each times for 3 times per week. The acupoints include SJ23 (Si Zhu Kong, unilateral), GB8 (Shuai Gu, unilateral), EX-HN5 (Tai Yang, unilateral), GB20 (Feng Chi, unilateral), LI4 (He Gu, bilateral), GB41 (Zu Lin Qi, bilateral), GB34 (Yang Ling Quan, bilateral) and SJ5 (Wai Guan, bilateral).

SUMMARY:
This study recruits 30 subjects into three groups, including two experimental groups and one control group. The two experimental groups receive acupuncture treatment for 4 weeks and two times functional magnetic resonance imaging scans as well as clinical symptom assessments. The control group receive one scan without any intervention. The aim of this study is to find the whether the effect of acupuncture treatment have diversity among migraineurs with different disease course.

DETAILED DESCRIPTION:
This study recruits 10 patients with long course (> 5 years) without aura migraine, 10 patients with short course (< 5 years) without aura migraine and 10 healthy volunteers who meet the inclusion and exclusion criteria. Among the study, two migraine patient groups receive acupuncture treatment for 4 weeks, the frequency is 30 minutes each time, three times a week. According to the national standard of the people's Republic of China (GB / T 12346-2006) acupoint name and location, the acupuncture treatment includes SJ23 (Si Zhu Kong, unilateral), GB8 (Shuai Gu, unilateral), EX-HN5 (Tai Yang, unilateral), GB20 (Feng Chi, unilateral), LI4 (He Gu, bilateral), GB41 (Zu Lin Qi, bilateral), GB34 (Yang Ling Quan, bilateral) and SJ5 (Wai Guan, bilateral) acupoints. Both migraine patients receive scan in functional magnetic resonance imaging (Siemens 3.0T superconducting magnetic resonance scanner, Germany) and symptom scale assessment before the first acupuncture stimulation and post the last acupuncture stimulation. Healthy volunteers receive only one scanning without intervention.

ELIGIBILITY:
Inclusion Criteria:

* Fitting to the standard of migraine without aura in the international classification of headache disease (ICHD-2) issued by the international headache society in 2004.
* Age from 18 to 55, male or female, with right-handedness.
* Having no depression or other serious mental illness.
* Having no psychoactive drugs taken in the past 3 months, or vasoactive drugs in the past 2 weeks.
* Having no habit of taking analgesics from a long time.

Exclusion Criteria:

* Having the first headache attack of migraine after 55 years old.
* Having a history of head injury, cluster headache, or other unclassified headaches.
* Taking medicine to prevent migraine in recent 4 weeks.
* Having the serious asymmetry or definite pathological changes in the anatomical structure of the head through the MRI scan.
* Cannot hold on the times of the MRI scan.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Headache Intensity | Change from Visual Analogue Scale at 1 months.
  The headache intensity is measured by the value of Visual Analogue Scale which limits 1 to 10. The higher value of this scale represents the worse headache.
Headache Days | Change from the number of day at 1 months.
  The days when headache attacked. The increased day represents the worse headache.
Headache Frequency | Change from the times of headache attack at 1 months.
  The maximum times in one day during the headache attacked. The increased time represents the worse headache.
Dataset of functional magnetic resonance imaging on brain | Changes from the dataset of subject's brain area at 1 months.
  Dataset of functional magnetic resonance imaging on brain includes functional images, structural images and diffusion tensor images.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Change from the value of Pittsburgh Sleep Quality Index at 1 months.
  One of the clinical measurement. The higher value represents the worse quality of sleep.
Medical Outcomes Study Short-Form 36 questionnaire | Change from the value of Medical Outcomes Study Short-Form 36 questionnaire at 1 months.
  One of the clinical measurement. The value range is 0 to 10, the higher value represents the better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ren, Doctor, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
The data of this study includes two aspect, data of brain scans and data of clinical symptom scales. The latter data will be shared to other researchers who contact us via email. The former data, however, is a DICOM format data that hard to analysis in non specialists. Besides, the size of DICOM data is much big that we haven't enough funding to support it in website. Thus, we haven't decided to share this kind of dataset. Except for those data, other data within our study is willing to be share.
  Our email: clancy_wu@bucm.edu.cn; clancy_wu@126.com; clancy.wu94@gmail.com.